CLINICAL TRIAL: NCT01075568
Title: The Satiety Effect After Okara Compared to Porridge Eating
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Nutrigal LTD (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: TASMC-10-NV-016-CTIL
Record Dates: First submitted 2010-02-17; First posted 2010-02-25 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-02

CONDITIONS: Healthy People

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Nutrigal Okara - 100

SUMMARY:
To examine the satiety effect after eating of Okara.

DETAILED DESCRIPTION:
This will be a single blind, cross-over design. Study population will include 10 subjects. The patients will be randomly assigned to receive one of two meals, 48 gram Okara or 40 gram (similar caloric value) semolina in two occasions (two visits). After the eating, the subject will stay in a closed room, without watch or any irritation. After three hours, the patient will fill a VAS questionnaire, and will get a standard meal. The meal will be weighed before and after.

Okara is a natural water extracted food grade soy product, contains approximately 35% protein (mfb), and about 43% of dietary fibers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 20-65 years old
* Written Informed Consent

Exclusion Criteria:

* History of gastro-intestinal surgery
* On medication that may influence gastric emptying, or medication for weight loss
* Patient on PPI treatment, H2 Blockers or medication for weight loss
* Known allergies to soy
* Pregnancy or breast-feeding
* Smoking
* Athletes
* Metabolic syndrome or diabetes mellitus
* Family history of metabolic syndrome or diabetes mellitus
* Weight loss > 2 kg during two months before the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To examine the satiety effect after 48 gram Okara compared to 40 gram of porridge eating.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel